CLINICAL TRIAL: NCT00239759
Title: Genetic Epidemiological Studies of Apolipoprotein E and Alzheimer's Disease
Brief Title: MIRAGE: Multi-Institutional Research in Alzheimer's Genetic Epidemiology
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Other Study IDs: IA0085; 2R01AG0902911-A2
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Alzheimer's Disease
Keywords: Epidemiological study
MeSH Terms: conditions — Alzheimer Disease

SUMMARY:
The goal of MIRAGE is to evaluate the association of genetic and non-genetic risk factors for Alzheimer's Disease.

DETAILED DESCRIPTION:
For the past 13 years the MIRAGE project has demonstrated that genetic factors play a major role in the development of Alzheimer's Disease (AD) among patients ascertained in clinical settings. This research has also shown that the E4 variant of apolipoprotein E (APOE), is the strongest AD risk factor identified thus far.

The researchers are turning their attention to the growing body of evidence from pathological, epidemiological and genetic studies that risk factors for vascular disease also enhance the risk of AD. However, since most epidemiological studies lack neuroimaging data, it is unclear whether the apparent association between vascular risk factors and AD is brought about by ischemic injury to the brain, acceleration of the primary Alzheimer neurodegenerative process, or some other process.

Some vascular risk factors are more prevalent in African American and Japanese American populations than in Caucasians. This study will build upon earlier work by evaluating the association between APOE, genes involved in vascular function, and other indictors of cerebrovascular health including blood pressure and structural brain imaging (MRI), and susceptibility to AD in these ethnic groups.

In order to carry out this project successfully, a sample of 1000 patients (500 Caucasians, 300 African Americans, 200 Japanese Americans) who meet NINCDS/ADRDA criteria for probable or definite AD from 11 centers in the U.S., Canada and Germany will be recruited. Many patients will be identified from the existing family registries. Family history, medical history, and epidemiological information will be obtained from the AD patient and their first-degree relatives using standardized questionnaire instruments and established protocols. A cognitive screening test will be administered to and blood samples will be collected from the patient's living siblings, spouses and children over the age of 50 years. DNA, plasma and MRI of the brain will be evaluated in patients and siblings.

ELIGIBILITY:
Inclusion Criteria:

NOTE: This trial accepts patients with Probable AD, and their cognitively normal brothers or sisters

* Probable or definite AD by NINCDS-ADRDA criteria
* Living siblings who are cognitively normal as measured by a brief standardized cognitive assessment
* Ages 60 and over for Alzheimer's disease patients
* Ages 50 and over for cognitively normal siblings

Exclusion Criteria:

* Early onset Alzheimer's disease attributed to APP, PS1 or PS2 gene mutations
* History of clinical stroke
* Siblings whose cognitive assessment does not meet study criteria
* Pacemaker or other contraindication to MRI

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2002-09; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Farrer, PhD, Principal Investigator — Chief, Genetics Program, Boston University
Locations (15):
- United States (12):
  - University of Alabama, Birmingham, Alabama
  - Sun Health Research Institute, Sun City, Arizona
  - Rancho Los Amigos National Rehabilitation Center/University of Southern California, Downey, California
  - University of California, Davis, Sacramento, California
  - Howard University, Washington D.C., District of Columbia
  - University of Miami School of Medicine, Miami Beach, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - Pacific Health Research Institute, Honolulu, Hawaii
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Boston University School of Medicine, Boston, Massachusetts
  - Cornell Medical University, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
- University of British Columbia, Vancouver, British Columbia, Canada
- Technical University of Munich, Munich, Germany
- G. Papanicolaou Hospital, Exholi Thessaloniki, Greece

REFERENCES:
- [Background] Bachman DL, Green RC, Benke KS, Cupples LA, Farrer LA; MIRAGE Study Group. Comparison of Alzheimer's disease risk factors in white and African American families. Neurology. 2003 Apr 22;60(8):1372-4. doi: 10.1212/01.wnl.0000058751.43033.4d. PMID 12707449
- [Background] Green RC, Cupples LA, Kurz A, Auerbach S, Go R, Sadovnick D, Duara R, Kukull WA, Chui H, Edeki T, Griffith PA, Friedland RP, Bachman D, Farrer L. Depression as a risk factor for Alzheimer disease: the MIRAGE Study. Arch Neurol. 2003 May;60(5):753-9. doi: 10.1001/archneur.60.5.753. PMID 12756140
- [Background] Henderson VW, Benke KS, Green RC, Cupples LA, Farrer LA; MIRAGE Study Group. Postmenopausal hormone therapy and Alzheimer's disease risk: interaction with age. J Neurol Neurosurg Psychiatry. 2005 Jan;76(1):103-5. doi: 10.1136/jnnp.2003.024927. PMID 15608005
- [Background] Yip AG, Green RC, Huyck M, Cupples LA, Farrer LA; MIRAGE Study Group. Nonsteroidal anti-inflammatory drug use and Alzheimer's disease risk: the MIRAGE Study. BMC Geriatr. 2005 Jan 12;5:2. doi: 10.1186/1471-2318-5-2. PMID 15647106
- [Background] Yip AG, McKee AC, Green RC, Wells J, Young H, Cupples LA, Farrer LA. APOE, vascular pathology, and the AD brain. Neurology. 2005 Jul 26;65(2):259-65. doi: 10.1212/01.wnl.0000168863.49053.4d. PMID 16043796
- See also: Boston University Alzheimer's Disease Center — http://www.bu.edu/alzresearch/